CLINICAL TRIAL: NCT05723757
Title: Autophagy Dysfunction in Hidradenitis Suppurativa
Acronym: AUTOPH-HS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Association pour la Recherche Clinique et Immunologique (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A01516-37
Record Dates: First submitted 2023-02-01; First posted 2023-02-13 (Actual); Last update posted 2023-02-13 (Actual); Status verified 2023-02

CONDITIONS: Hidradenitis Suppurativa (HS)
MeSH Terms: conditions — Hidradenitis Suppurativa | interventions — Blood Specimen Collection

STUDY DESIGN:
Intervention Model Description: This is an exploratory, intra-individual, prospective, mono-site study. This study is a category 2 study (interventional research with minimal risks and constraints).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- HS Patients (Experimental): 50 adult subjects suffering from moderate to severe HS, aged 18 to 65, diagnosed for at least 1 year
  Interventions: Diagnostic Test: blood sampling

INTERVENTIONS:
Diagnostic Test: blood sampling — Draw a 8.5mL blood sample for detection of SNPs of genomic origin

SUMMARY:
The pathogenesis of HS is still poorly understood: the pilosebaceous tropism and the fact that patients respond to combinations of antibiotics and/or immunosuppressive treatments suggest the involvement of 3 factors that would be intimately linked: the presence of (i) a microbial dysbiosis, (ii) a dysfunction of the pilosebaceous apparatus and (iii) an inappropriate immune response. But how these 3 elements interact with each other remains unestablished, with few studies that have analyzed them from a kinetic point of view. Beyond a possible dysfunction of the pilosebaceous apparatus, we hypothesize a bacterial dysbiosis in connection with abnormalities of autophagy function with secondary development of an inappropriate immune response. Because of its functions of bacterial clearance and activation of local immune response, a defect in the autophagic process may be associated with the development of inflammatory pathologies related to microbial dysbiosis. Crohn's disease (CD), an inflammatory pathology of the gastrointestinal tract associated with intestinal dysbiosis, has been associated with alterations in autophagy, with approximately 50% of patients having single nucleotide polymorphisms (SNPs) associated with autophagy deficiency (Ellinghaus et al., 2013). The epidemiological association of CD/HS, the presence of skin dysbiosis and a chronic inflammatory response during HS, make us suspect a deficit of autophagic function in these patients, in a similar way to what is observed during Crohn's disease.

The aim of this study is to analyze the frequency of 100 SNPs, reported to be associated with autophagy deficiency, in a cohort of moderate-to-severe HS patients.

ELIGIBILITY:
Inclusion Criteria:

* Subject aged 18 to 65 years (included)
* Subject diagnosed with HS for at least 1 year
* Subject diagnosed with moderate-to-severe HS defined by HS PGA≥3
* Subject presenting an HS with inflammatory phenotype defined by the presence of folliculitis, nodules and/or abcesses
* Subject suffering from at least 4 flares/year and presenting 5 active inflammatory lesions (nodules and/or abcesses)
* Subject able to read, understand and give documented informed consent
* Subject willing and able to comply with the protocol requirements for the duration of the study
* Subject with health insurance coverage according to local regulations

Exclusion Criteria:

* - Pregnancy or breast-feeding women
* Subject currently experiencing or having a history of other concomitant skin or systemic inflammatory conditions that could constitute a bias (i.e. psoriasis, Crohn's Disease, etc.)
* Subject with any additional condition that, in the opinion of the investigator, may interfere with the assessment or put the subject at risk
* Linguistic or mentally incapacity to sign the consent form
* Subject protect by the law (adult under guardianship, or hospitalized in a public or private institution for a reason other than study, or incarcerated)
* Subject in an exclusion period from a previous study or who is participating in another clinical trial using a drug

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Prevalence of 100 SNPs in genomic DNA (blood) associated with autophagy deficiency | Day 0
  Prevalence of 100 SNPs in genomic DNA (blood) associated with autophagy deficiency in a cohort of moderate-to-severe HS patients The prevalence of these SNPs will be compared with the prevalence observed in a population suffering from Crohn's Diseases (Ellinghaus et al., 2013).

SECONDARY OUTCOMES:
Prevalence of 100 SNPs in somatic DNA (skin) associated with autophagy deficiency in a cohort of moderate-to-severe HS patients | Day 0
  The prevalence of these SNPs will be compared with the prevalence of SNPs in genomic DNA (blood) Prevalence of 100 SNPs associated with autophagy deficiency in genomic DNA (blood) and somatic DNA (skin)
Prevalence of 100 SNPs in genomic DNA (blood) and somatic DNA (Skin) associated with autophagy deficiency according to severity of disease. | Day 0
  Prevalence of 100 SNPs in genomic DNA (blood) associated with autophagy deficiency according to severity of disease. The severity of HS disease will be evaluated through clinical scores (HS PGA scale, IH-S4 score, Hurley stage or refined Hurley) or quality of life score (DLQI). Prevalence of 100 SNPs in somatic DNA (skin) associated with autophagy deficiency according to severity of disease. The severity of HS disease will be evaluated through clinical scores (HS PGA scale, IH-S4 score, Hurley stage or refined Hurley) or quality of life score (DLQI). Prevalence of 100 SNPs associated with autophagy deficiency in genomic DNA (blood) and somatic DNA (skin), according to severity of disease. The severity of HS disease will be evaluated through clinical scores (HS PGA scale, IH-S4 score, Hurley stage or refined Hurley) or quality of life score (DLQI).

IPD SHARING:
Plan to Share IPD: No